CLINICAL TRIAL: NCT01681004
Title: INSITE Investigation of Sacroiliac Fusion Treatment
Brief Title: Investigation of Sacroiliac Fusion Treatment (INSITE)
Acronym: INSITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300103
Record Dates: First submitted 2012-09-01; First posted 2012-09-07 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Degenerative Sacroiliitis; Sacroiliac Joint Disruption
Keywords: si joint; si joint pain; si joint injury; si joint treatment; si joint injections; si joint inflammation; si joint problems; si joint symptoms; hypermobile si joint; si joint arthritis; si joint pain treatment; inflamed si joint; si joint sclerosis; locked si joint; si joint injuries; si joint disease; si joint infection; sacroiliac joint pelvic pain; sacroiliac joint arthritis treatment

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- iFuse Implant System (Experimental): Surgical placement of iFuse implants in the affected SI joint
  Interventions: Device: iFuse Implant System
- Non-Surgical Management (Active Comparator): Medications, SI joint injection, physical therapy and RF ablation of SI joint
  Interventions: Other: Non-surgical management

INTERVENTIONS:
Device: iFuse Implant System — Placement of iFuse implant system via surgery
  Arms: iFuse Implant System
Other: Non-surgical management — Medications for pain, physical therapy, SI joint injection and RF ablation
  Arms: Non-Surgical Management

SUMMARY:
The purpose of this study is to compare outcomes when patients with degenerative sacroiliitis (arthritis of the SI joint) and or sacroiliac disruption (abnormal separation or tearing of the sacroiliac joint)undergo either SI joint fusion with the iFuse Implant System or undergo specific, targeted non-surgical treatment of the SI joint.

DETAILED DESCRIPTION:
The intended analysis was to examine differences in responses at 6 months. It was acknowledged that subjects with chronic pain in the NSM arm group might not experience any benefit as there was little evidence at the time that NSM was helpful. The protocol included optional crossover to other treatments, including surgical treatment. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 at time of screening
2. Patient has lower back pain for >6 months inadequately responsive to conservative care
3. Diagnosis of sacroiliac joint disruption or degenerative sacroiliitis based on ALL of the following:

   1. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test), and
   2. Patient has at least 3 of 5 physical examination maneuvers specific for the SI joint (see Table 3), and
   3. Patient has improvement in lower back pain numeric rating scale (NRS) of at least 50% after injection of local anesthetic into affected SI joint(s) (see Section 3.6.4), and
   4. One or more of the following:

   i. SI joint disruption:
   * Asymmetric SI joint widening on X-ray or CT scan, or
   * Leakage of contrast on diagnostic arthrography

   ii. Degenerative sacroiliitis:
   * Radiographic evidence of SI joint degeneration, including sclerosis, osteophytes, subchondral cysts, or vacuum phenomenon on CT or plain film, or
   * Due to prior lumbosacral spine fusion
4. Baseline Oswestry Disability Index (ODI) score of at least 30%
5. Baseline SI joint pain score of at least 50 on 0-100 mm visual analog scale*
6. Patient has signed study-specific informed consent form
7. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements

Exclusion Criteria:

1. Severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture**
2. Other known sacroiliac pathology such as:

   1. Sacral dysplasia
   2. Inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondyloarthropathy)
   3. Tumor
   4. Infection
   5. Acute fracture
   6. Crystal arthropathy
3. History of recent (<1 year) major trauma to pelvis
4. Previously diagnosed osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture). Patients meeting the osteoporosis screening criteria identified by the National Osteoporosis Foundation should be screened for osteoporosis with DEXA.**** See Section 3.6.4.
5. Osteomalacia or other metabolic bone disease
6. Chronic rheumatologic condition (e.g., rheumatoid arthritis)
7. Any condition or anatomy that makes treatment with the iFuse Implant System infeasible
8. Chondropathy
9. Known allergy to titanium or titanium alloys
10. Use of medications known to have detrimental effects on bone quality and soft-tissue healing
11. Prominent neurologic condition that would interfere with physical therapy
12. Current local or systemic infection that raises the risk of surgery
13. Patient currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation.
14. Currently pregnant or planning pregnancy in the next 2 years
15. Patient is a prisoner or a ward of the state.
16. Known or suspected drug or alcohol abuse***
17. Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
18. Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cher, MD, Principal Investigator — SI-BONE
Locations (19):
- United States (19):
  - University of California, San Diego, La Jolla, California
  - BASIC Spine, Newport Beach, California
  - University of Colorado Denver Health Sciences, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Orthopaedic Clinic of Daytona Beach, Daytona Beach, Florida
  - Brain and Spine Center, LLC, Panama City, Florida
  - Resurgen's Orthopaedics, McDonough, Georgia
  - Neurosurgery Consultants/ Riverside Hospital, Kankakee, Illinois
  - Orthopaedic Center of Southern Illinois, Mount Vernon, Illinois
  - Community Neurosurgery Hospital, Indianapolis, Indiana
  - Bluegrass Orthopaedics & Hand Care Research, Lexington, Kentucky
  - Spine institute of Louisiana, Shreveport, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - HCA Midwest, Kansas City, Missouri
  - NeuroSpine Institute, LLC, Eugene, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Midwest Orthopedic Specialty Hospital, Franklin, Wisconsin
  - Aurora Bay Care Medical Center, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Polly DW, Swofford J, Whang PG, Frank CJ, Glaser JA, Limoni RP, Cher DJ, Wine KD, Sembrano JN; INSITE Study Group. Two-Year Outcomes from a Randomized Controlled Trial of Minimally Invasive Sacroiliac Joint Fusion vs. Non-Surgical Management for Sacroiliac Joint Dysfunction. Int J Spine Surg. 2016 Aug 23;10:28. doi: 10.14444/3028. eCollection 2016. PMID 27652199
- [Result] Polly D, Cher D, Whang PG, Frank C, Sembrano J; INSITE Study Group. Does Level of Response to SI Joint Block Predict Response to SI Joint Fusion? Int J Spine Surg. 2016 Jan 21;10:4. doi: 10.14444/3004. eCollection 2016. PMID 26913224
- [Result] Cher DJ, Frasco MA, Arnold RJ, Polly DW. Cost-effectiveness of minimally invasive sacroiliac joint fusion. Clinicoecon Outcomes Res. 2015 Dec 18;8:1-14. doi: 10.2147/CEOR.S94266. eCollection 2016. PMID 26719717
- [Result] Polly DW, Cher DJ, Wine KD, Whang PG, Frank CJ, Harvey CF, Lockstadt H, Glaser JA, Limoni RP, Sembrano JN; INSITE Study Group. Randomized Controlled Trial of Minimally Invasive Sacroiliac Joint Fusion Using Triangular Titanium Implants vs Nonsurgical Management for Sacroiliac Joint Dysfunction: 12-Month Outcomes. Neurosurgery. 2015 Nov;77(5):674-90; discussion 690-1. doi: 10.1227/NEU.0000000000000988. PMID 26291338
- [Result] Whang P, Cher D, Polly D, Frank C, Lockstadt H, Glaser J, Limoni R, Sembrano J. Sacroiliac Joint Fusion Using Triangular Titanium Implants vs. Non-Surgical Management: Six-Month Outcomes from a Prospective Randomized Controlled Trial. Int J Spine Surg. 2015 Mar 5;9:6. doi: 10.14444/2006. eCollection 2015. PMID 25785242
- Available data/document: Individual Participant Data Set: INSITE — http://yoda.yale.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 442 patients who were screened for participation at 19 sites, 159 (37.8%) were enrolled. Eleven subjects withdrew before treatment (1 before randomization and 10 after randomization but before any treatment was performed), yielding a total of 148 subjects who were enrolled, randomized and treated.
Groups:
- Non-Surgical Management: Medications, SI joint injection, physical therapy and RF ablation of SI joint
  Non-surgical management: Medications for pain, physical therapy, SI joint injection and RF ablation.
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
Period: Primary Endpoint: 6 Months
Arm/Group | iFuse Implant System | Non-Surgical Management
Started | 102 | 46
Crossover to Surgical Treatment | 0 | 39 (Crossover to surgical treatment allowed per study protocol after the 6-month visit was complete.)
Completed | 101 | 44
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Study Completion
Arm/Group | iFuse Implant System | Non-Surgical Management
Started | 101 | 44
Completed | 89 | 36
Not Completed | 12 | 8
Not completed — Lost to Follow-up | 8 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Site Termination | 2 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 442 patients who were screened for participation at 19 sites, 159 (37.8%) were enrolled. Eleven subjects withdrew before treatment (1 before randomization and 10 after randomization but before any treatment was performed), yielding a total of 148 subjects who were enrolled, randomized and treated (102 to iFuse Implant System & 46 to NSM).
Groups:
- Non-Surgical Management: Medications, SI joint injection, physical therapy and RF ablation of SI joint
  Non-surgical management: Medications for pain, physical therapy, SI joint injection and RF ablation
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
- Total: Total of all reporting groups
Arm/Group | iFuse Implant System | Non-Surgical Management | Total
Number analyzed (Participants) | 102 | 46 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 38 | 130
  >=65 years | 10 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 28 | 103
  Male | 27 | 18 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 97 | 44 | 141
  Black | 3 | 2 | 5
  American Indian | 1 | 0 | 1
  Other | 1 | 0 | 1
  Ethnicity: Hispanic or Latino | 4 | 4 | 8
Body Mass Index, mean (range) [Mean (Full Range); unit: kg / m2] | 30.4 [16.7 to 49.5] | 30.6 [19.4 to 48.9] | 30.43 [16.7 to 49.5]
Smoking Status (n, %) [Number; unit: participants]
  Current Smoker | 26 | 3 | 29
  Former Smoker | 30 | 13 | 43
  Never smoker | 46 | 30 | 76
Ambulatory without assistance [Count of Participants; unit: Participants] | 89 | 41 | 130
Work status (n, %) [Count of Participants; unit: Participants]
  Working full time | 45 | 21 | 66
  Working part time | 9 | 4 | 13
  Not working, student | 1 | 0 | 1
  Not working, retired | 21 | 9 | 30
  Not working due to back pain | 20 | 8 | 28
  Not working other reason | 6 | 4 | 10
Prior Lumbar fusion (n, %) [Count of Participants; unit: Participants] | 41 | 17 | 58
Underlying diagnosis [Count of Participants; unit: Participants]
  Degenerative sacroiliitis | 88 | 40 | 128
  Sacroiliac joint disruption | 14 | 6 | 20
Years of pain, mean (range) [Mean (Full Range); unit: years] | 7.0 [0.5 to 40.7] | 5.0 [0.5 to 38.9] | 6.0 [0.5 to 40.7]
Pain Syndrome [Count of Participants; unit: Participants]
  Pain began peripartum | 29 | 19 | 48
  Pain radiates down leg | 89 | 41 | 130
  Groin pain | 60 | 29 | 89
  Pain worse with sitting | 89 | 41 | 130
  Pain worse with rising | 88 | 41 | 129
  Pain worse with walking | 87 | 42 | 129
  Pain worse with climbing stairs | 93 | 41 | 134
  Pain worse with descending stairs | 82 | 37 | 119
Prior treatments [Count of Participants; unit: Participants]
  Physical therapy | 71 | 36 | 107
  Steroid SIJ injection | 85 | 42 | 127
  RF ablation | 21 | 4 | 25
Taking opiods [Count of Participants; unit: Participants] | 70 | 29 | 99
Participants with lumbar stenosis [Count of Participants; unit: Participants] | 15 | 7 | 22
Participants with hip diagnosis (n, %) [Count of Participants; unit: Participants] | 16 | 3 | 19
Participants with sacral trauma (n, %) [Count of Participants; unit: Participants] | 8 | 3 | 11
VAS SIJ pain score, mean [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Scale (VAS) is a 100 mm line on which the subjects mark their pain rating. 0= no pain and 100= worst pain imaginable.
  units on a scale | 82.3 (11.9) | 82.2 (9.9) | 82.3 (11.3)
ODI score, mean [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index is a validated measure of disability related to low back pain. There are 10 sections, each with a score between 0-5. If all sections are answered, the total possible score is 50/50 = 100% which is the worst disability possible on the scale. (0/50 = no disability at all.) If any section is skipped by the study participant, the total possible score for that section is removed from the denominator. Example - section 8 skipped, total possible score is 45/45 = 100%.
  units on a scale | 57.2 (12.8) | 56.0 (14.0) | 56.8 (13.2)
SF-36, mean [Mean (Standard Deviation); unit: units on a scale] — The Short Form 36 health survey (SF-36) is a 36-item patient reported health questionnaire to measure quality of life across 8 domains.
  The PCS is the Physical Component Summary score. 0% would represent the lowest or worst possible level of functioning while 100% would represent the highest / best possible level of functioning.
  The MCS is the Mental Component Summary score. 0% would represent the lowest or worst possible level of functioning while 100% would represent the highest / best possible level of functioning.
  units on a scale
    Physical component summary (PCS) | 30.2 (6.2) | 30.8 (6.2) | 30.4 (6.2)
    Mental component summary (MCS) | 43.0 (11.5) | 43.3 (12.1) | 43.1 (11.6)
EQ-5D [Mean (Standard Deviation); unit: units on a scale] — EQ-5D is a five-question broad quality of life measure that is combined into a single index using population norm data called time trade-off (TTO) utility of current health. A score of 0 would = worst imaginable health, while a score of 1.0 would be best imaginable health. (Scores <0 are also possible, representing states worse than death.) EQ-5D also includes a 0-100 mm health thermometer, where 0 means death and 100 means perfect health.
  units on a scale
    Time trade-off (TTO) score | 0.44 (0.18) | 0.47 (0.19) | 0.45 (0.18)
    Health Thermometer | 53.2 (23.8) | 57.8 (22.9) | 54.6 (23.5)

OUTCOME MEASURES:

1. Primary Outcome: Subject Success
Description: Composite endpoint of reduction from baseline in VAS back pain score by at least 20 mm, lack of device-related serious adverse events, absence of neurologic worsening and absence of surgical re-intervention. Note that the primary endpoint analysis is **intent to treat**, meaning that an outcome (success or failure) is assigned to all subjects randomized and treated. Subjects who withdrew early were deemed study failures.
Time Frame: 6 months
Population: A modified intent-to-treat approach was used.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Surgical Management: This arm includes all subjects randomized to NSM with reporting to 6 months only.
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 102 | 46
Participants | 84 | 12

2. Secondary Outcome: Improvement in SI Joint Pain VAS Score at 1 Month
Description: Improvement in SI joint pain VAS score of greater than or equal to 20 points, at post-operative & NSM visit after 1 month. The Visual Analog Scale (VAS) is a 100 mm line on which the subject indicates their level of pain. 0 = no pain. 100 = worst imaginable pain. Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 1 month
Population: 2 iFuse and 1 NSM subjects did not complete the pain score.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Surgical Management: This arm includes all subjects randomized to NSM.
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 45
Participants | 84 | 13

3. Secondary Outcome: Improvement in Si Joint Pain VAS Score at 3 Months
Description: Improvement in SI joint pain VAS score of greater than or equal to 20 points, at post-operative & NSM visits after 3 months. The Visual Analog Scale (VAS) is a 100 mm line on which the subject indicates their level of pain. 0 = no pain. 100 = worst imaginable pain. Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 3 Months
Population: 2 iFuse and 3 NSM subjects did not complete the 3-month pain score.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 43
Participants | 87 | 17

4. Secondary Outcome: Improvement in SI Joint Pain VAS Score at 6 Months
Description: Improvement in SI joint pain VAS score of greater than or equal to 20 points, at post-operative & NSM visits after 6 months. The Visual Analog Scale (VAS) is a 100 mm line on which the subject indicates their level of pain. 0 = no pain. 100 = worst imaginable pain. Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 6 Months
Population: 1 iFuse and 3 NSM subjects did not complete the 6-month pain score.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 101 | 43
Participants | 84 | 12

5. Secondary Outcome: Improvement in SI Joint Pain VAS Score at 12 Months
Description: Improvement in SI joint pain VAS score of greater than or equal to 20 points compared to baseline. The Visual Analog Scale (VAS) is a 100 mm line on which the subject indicates their level of pain. 0 = no pain. 100 = worst imaginable pain. Note that secondary endpoint analysis is based on available data only. Subjects in the NSM group who crossed over are considered failures for this endpoint by definition.
Time Frame: 12 Months
Population: 2 iFuse subjects did not complete the 12-month pain score. Analysis of 12-month scores in the NSM group is not valid because of the high crossover rate.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Surgical Management: This arm includes all subjects randomized to NSM followed to 6 months.
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 6
Participants | 81 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

6. Secondary Outcome: Improvement in SI Joint Pain VAS Score at 24 Months
Description: as for outcome 5
Time Frame: 24 Months
Population: 12 iFuse subjects did not complete the 24-month pain score. Analysis of 24-month scores in the NSM group is not valid because of the high crossover rate.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 90 | 5
Participants | 75 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

7. Secondary Outcome: Improvement in Back Dysfunction
Description: Improvement in ODI score of greater than or equal to 15 points, at month 1.
  Oswestry Disability Index is a validated measure of disability related to low back pain. There are 10 sections, each with a score between 0-5. Scores are expressed on a percent basis without using the percent term. Scores range from 0 (no disability) to 100 (completely disabled).
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 1 month
Population: 2 iFuse and 1 NSM subjects did not complete ODI at 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 45
Participants | 49 | 6

8. Secondary Outcome: Improvement in Back Dysfunction
Description: Improvement in ODI score of greater than or equal to 15 points, at month 3.
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 3 Months
Population: 2 iFuse subjects and 3 NSM subjects did not complete ODI at month 3.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 43
Participants | 72 | 13

9. Secondary Outcome: Improvement in Back Dysfunction
Description: Improvement in ODI score of greater than or equal to 15 points, at post-operative visits. 6 month visit.
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 6 Months
Population: 1 iFuse and 2 NSM subjects did not complete ODI at month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 101 | 44
Participants | 74 | 6

10. Secondary Outcome: Improvement in Back Dysfunction
Description: Improvement in ODI score of greater than or equal to 15 points compared to baseline. Oswestry Disability Index is a validated measure of disability related to low back pain. Subjects in the NSM group who crossed over are considered failures for this endpoint by definition.
Time Frame: 12 Months
Population: 2 iFuse subjects did not complete ODI at month 12. ODI analysis is not valid in NSM group at 12 months because of high crossover.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 6
Participants | 72 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

11. Secondary Outcome: Improvement in Back Dysfunction
Description: as for outcome 10
Time Frame: 24 Months
Population: The Count of participants = number of subjects that had a threshold change in ODI score of greater than or equal to 15 points. Overall number of participants = number of subjects analyzed. Of the 102, a total of 13 iFuse Implant subjects exited the study and 1 did not complete the ODI survey. By 6 months, 39 NSM subjects crossed over to surgical.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 88 | 40
Participants | 60 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

12. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by SF-36 PCS (Physical Component) at Post-operative Visits
Description: Improvement in quality of life (QOL) as measured by SF-36 PCS (Physical Component) at post-operative / NSM visits. The Short Form 36 health survey (SF-36) is a 36-item patient reported health questionnaire to measure quality of life across 8 domains. The PCS is the Physical Component Summary score. PCS is normed, so that "normal" scores are 50 +- 10. Higher scores indicate higher quality of life; lower scores indicate lower quality of life. SF-36 PCS (NBS, 2009 norms) ranges from 5 (minimum value, poor physical function) to 80 (maximum, excellent clinical function).
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 6 months
Population: 2 iFuse and 2 NSM subjects did not complete SF-36 at month 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 44
units on a scale | 12.5 (10.5) | 1.3 (8.2)

13. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by SF-36 PCS (Physical Component) at Post-operative Visits
Description: as for outcome 12
Time Frame: 12 Months
Population: A total of 2 iFuse subjects had exited the study before making it to their 12 month visit. This outcome is not evaluated in the NSM group at month 12 because high crossover to surgical treatment prevents valid analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 6
units on a scale | 13.0 (9.9) | NA (NA) — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

14. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by SF-36 PCS (Physical Component) at Post-operative Visits
Description: as for outcome 12
Time Frame: 24 months
Population: Change in QOL score at 24 months. 89 participants had QOL information at 24 months. Analysis of the NSM cohort is not done because high crossover to surgery prevents valid analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 89 | 5
units on a scale | 11.2 (10.7) | NA (NA) — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

15. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by EQ-5D (EuroQol-5D) at Post-operative Visits
Description: Improvement in quality of life (QOL) as measured by EQ-5D (EuroQol-5D) at post-operative visits. EQ-5D is a five-question broad quality of life measure that can be combined into a single index and represents the time trade-off (TTO) utility of current health. A score of 0 would = worst imaginable health, while a score of 1.0 would be best imaginable health.
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 6 months
Population: Results show improvement in score from baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 44
units on a scale | 0.29 (0.22) | 0.06 (0.28)

16. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by EQ-5D (EuroQol-5D) at Post-operative Visits
Description: as for outcome 15
Time Frame: 12 Months
Population: 2 iFuse subjects did not complete the survey at month 12. Due to high crossover rate to surgery, analysis in the NSM group is not valid.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 100 | 6
units on a scale | 0.31 (0.22) | NA (NA) — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

17. Secondary Outcome: Improvement in Quality of Life (QOL) as Measured by EQ-5D (EuroQol-5D) at Post-operative Visits
Description: as for outcome 15
Time Frame: 24 months
Population: 13 iFuse subjects did not complete the 24-month assessment. Analysis was not done for the NSM group at 24 months due to the high crossover rate.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 89 | 5
units on a scale | 0.29 (0.24) | NA (NA) — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

18. Secondary Outcome: Ambulatory Status
Description: Time to full ambulation among those without full ambulation at baseline.
  60 days was the median of time to full ambulation for the iFuse implant System arm.
Time Frame: 24 months (surgical group), 6 months (non-surgical group)
Population: Number of days to full ambulation among those without full ambulation at baseline. At baseline only 13 in the surgical arm were not Ambulatory without assistance and for the NSM group, it was only 5 at baseline.
Measure: Median (95% Confidence Interval); unit: Days, median
Groups:
- Non-Surgical Management: This arm includes all subjects randomized to NSM followed to 6 months..
  Subjects were allowed to cross over to other treatments (including surgical treatments) after the month 6 visit was complete.
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 13 | 5
Days, median | 60 [46 to NA] — Upper confidence limit not defined due to small sample size. | NA [NA to NA] — By month 6, only 40% of non-ambulatory NSM subjects regained full ambulation status

19. Secondary Outcome: Work Status
Description: Proportion of non-working (due to back pain or other reasons) subjects who return to work
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 1 month
Population: Patients not working at baseline due to back or other pain. Note this is a subset of the entire population.
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 26 | 12
Participants | 2 | 0

20. Secondary Outcome: Work Status
Description: Non-working subjects (due to back pain or other reasons) who return to work
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 3 Months
Population: Patients not working at baseline due to back or other pain
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 26 | 12
Participants | 3 | 0

21. Secondary Outcome: Work Status
Description: Non-working subjects who return to work
  Note that secondary endpoint analysis is based on available data only. No imputation of missing scores was prespecified in the protocol.
Time Frame: 6 Months
Population: Patients not working at baseline due to back or other pain
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 26 | 12
Participants | 5 | 0

22. Secondary Outcome: Work Status
Description: as for outcome 21
Time Frame: 12 Months
Population: Patients not working at baseline due to back or other pain
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 26 | 6
Participants | 4 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

23. Secondary Outcome: Work Status
Description: as for outcome 21
Time Frame: 18 Months
Population: Patients not working at baseline due to back or other pain
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 23 | 5
Participants | 3 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

24. Secondary Outcome: Work Status
Description: as for outcome 21
Time Frame: 24 Months
Population: Patients not working at baseline due to back or other pain
Measure: Count of Participants; unit: Participants
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 23 | 5
Participants | 2 | NA — The intended analysis was to examine differences in responses at 6 months. The protocol anticipated a high crossover rate and therefore did not include any comparative analyses after month 6.

25. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Any event meeting ISO 14155 definition for serious adverse event at following time points: during procedure (if randomized to iFuse), hospital discharge (if iFuse, typically 1-2 days), and 1, 3, 6, 12, 18 and 24 months after randomization.
Time Frame: Procedure, discharge, 1, 3, 6, 12, 18 and 24 months
Population: All treated study subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Surgical Management: This arm includes all subjects randomized to NSM. Many of these subjects crossed over to treatment after 6 months of NSM.
Arm/Group | iFuse Implant System | Non-Surgical Management
Number analyzed (Participants) | 102 | 46
Participants | 38 | 12

ADVERSE EVENTS:
Time Frame: 1 month, 3 months, 6 months, 12 months, 18 months, 24 months
Groups:
- iFuse Implant System: Surgical placement of iFuse implants in the affected SI joint iFuse Implant System: Placement of iFuse implant system via surgery
- Non-Surgical Management: This arm includes all subjects randomized to NSM followed to 6 months
  Non-surgical management: Medications for pain, physical therapy, SI joint injection and RF ablation.
Arm/Group | iFuse Implant System | Non-Surgical Management
All-Cause Mortality (participants affected / at risk) | 1/102 | 1/46
Serious Adverse Events (participants affected / at risk) | 38/102 | 12/46
Other Adverse Events (participants affected / at risk) | 69/102 | 35/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iFuse Implant System (N=102) | Non-Surgical Management (N=46)
Osteoarthritis of the knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meniscal tear (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Contralateral SIJ pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
Degenerative disease - spine (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Disc herniation (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Ipsilateral - SIJ pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis of the hip (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Avascular necrosis of left hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Restrolisthesis T12-L1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture - tibia / fibula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Labral tear & ilium fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Snapping scapula syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wound hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Revision - SIJ pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Revision - neuropathy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neuropathy - Resolved with revision (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation / respira failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction - fatal (Cardiac disorders) | 1 (1) | 0 (0) — Myocardial infarction - fatal
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruct, leading to surgery (Gastrointestinal disorders) | 1 (1) | 0 (0) — Bowel obstruct, leading to surgery
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
S1 neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Benign prostatic hypertrophy (General disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kidney disfunction due to nsaid (Renal and urinary disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iFuse Implant System (N=102) | Non-Surgical Management (N=46)
Knee pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (29) | 8 (8)
Degenerative disease - spine (Musculoskeletal and connective tissue disorders) | 17 (19) | 12 (16)
SIJ pain - ipsilateral (Musculoskeletal and connective tissue disorders) | 13 (14) | 10 (11)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
SIJ pain - contralateral (Musculoskeletal and connective tissue disorders) | 12 (12) | 6 (6)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 12 (14) | 4 (4)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Hip pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Upper respiratory infection (Infections and infestations) | 5 (5) | 4 (5)

LIMITATIONS AND CAVEATS:
Open-label (non-blinded) study. Most (>90%) NSM subjects with continued pain crossed over after the 6-month visit. Analysis across groups after 6 months is therefore biased, since surgery by definition is not a component of non-surgical treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No